CLINICAL TRIAL: NCT04486131
Title: Lateral Nodal Recurrence in Rectal Cancer
Acronym: LaNoReC
Status: Recruiting | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, M. Kusters, Principal Investigator, Amsterdam UMC, location VUmc
Other Study IDs: A2021.0524.0001
Record Dates: First submitted 2020-06-30; First posted 2020-07-24 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Local recurrence rates in rectal cancer have reduced dramatically since the introduction of the total mesorectal excision (TME) technique and neoadjuvant (chemo)radiotherapy (C))RT) to overall rates of 5-year local recurrence to 5-10%.

However, distal rectal cancers have a tendency to spread to lateral lymph nodes and it was recently shown that patients with enlarged lateral lymph nodes of ≥7mm short-axis size have a considerable chance of a local recurrence: 15-20%. This is regardless of CRT with TME in two retrospective cohorts (Lateral Node Consortium and Snapshot Rectal Cancer 2016 study). According to the Lateral Node Consortium study, this rate was significantly reduced to <6% when performing a lateral lymph node dissection (LLND) after (C)RT + TME.

A major drawback of these recent multi-center studies is their retrospective nature. Therefore, in the Netherlands, radiologists, radiation oncologists, surgeons and pathologists have recently been educated and trained to enhance knowledge and awareness of LLNs and to implement nerve-sparing minimally invasive LLND.

The LaNoReC trial is a prospective registration study aimed at evaluating oncological outcomes after multi-disciplinary training. The main question of this study is whether, after dedicated training and the performance of LLNDs, the lateral local recurrence rate in rectal cancers with enlarged nodes (≥7mm) can be reduced to below 6%.

DETAILED DESCRIPTION:
Local recurrence rates in rectal cancer have reduced dramatically since the introduction of the total mesorectal excision (TME) technique. These rates have been lowered further with the use of neoadjuvant (chemo)radiotherapy ((C)RT) regimens in appropriate cases, decreasing overall rates of 5-year local recurrence to 5-10%. However, in patients with enlarged lateral lymph nodes (LLNs, ≥7mm short-axis size), recurrence rates have remained high, up to 20%. Most likely, this is caused by lymphatic spread of low rectal cancer to the lateral compartments. Western surgeons have always relied on (C)RT to sterilize the lateral compartments, containing the internal iliac and obturator lymph nodes, alleviating fears of operative morbidity and nerve function disorders associated with a lateral lymph node dissection (LLND), mainly performed in the East. Furthermore, most Western clinicians consider lateral nodal disease to represent metastatic disease, not amendable to cure.

The Lateral Node Consortium undertook a multi-centre study with 12 centres from seven countries, collecting data over a 5-year period, including all consecutive patients operated for a cT3 or T4 rectal cancer. In all patients, every series of MRIs was re-reviewed by a standardized protocol, examining lateral pelvic nodes, defining these according to size and the presence of malignant features and relating these to the development of locally recurrent disease. In the first publication of the consortium with a total of 1216 patients, it was shown that pre-treatment lateral lymph node (LLN) size of ≥7 mm, results in an unacceptably high incidence of lateral local recurrence of 20%, despite (C)RT with TME. Within the consortium, several centres performed LLND's after (C)RT, which resulted in a significantly lower rate of lateral local recurrence of 6% in nodes ≥7 mm (p = 0.042). Furthermore, LLN enlargement did not influence distant metastases rate, suggesting it is a local issue which requires to be addressed through targeted treatment in the pelvis, rather simply representing a marker of poor prognosis and distant disease.

Additionally, a second study, the Snapshot Rectal Cancer 2016 was conducted in 2020. This national retrospective cohort study included 3057 patients operated for rectal cancer in 2016 with a 4-year follow-up period. Radiologists were trained for LLN classification and measurements and re-reviewed MRIs of 882 patients with low (≤8cm from the anorectal junction), cT3/4 rectal cancer who received neoadjuvant (chemo)radiotherapy with the help of two atlases. This study found a 4-year LLR risk of 15% in presence of enlarged LLNs.

The major drawback of these multi-center studies are their retrospective nature. Radiological reporting of LLNs was low for primary MRIs, which may have influenced treatment decisions. Consequently, LLNs may have not been separately included in irradiation field. Moreover, neither study was able to investigate the effect of LLND in a trained setting. In the Netherlands, radiologists, radiation oncologists, surgeons and pathologists have recently been educated and trained to enhance knowledge and awareness of LLNs and to implement nerve-sparing minimally invasive LLND. The LaNoReC describes a prospective evaluation of oncological outcomes after multi-disciplinary training, thereby aiming for a 50% reduction in LLR rates.

ELIGIBILITY:
Inclusion Criteria:

• All patients with rectal cancer with one or more lateral nodes with a short-axis of ≥7mm or ≥5mm with one or more malignant features (i.e. round shape, irregular margins, heterogeneity, loss of fatty hilum).

Exclusion Criteria:

* Younger than 18 years old
* Pelvic irradiation in the medical history
* Previous lateral lymph node dissection related to pelvic malignancy
* Synchronous distant metastases
* Familiar adenomatous polyposis
* Synchronous colon cancer with a higher stage than rectal cancer
* Absolute contraindication for general anaesthesia
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rectal cancer with one or more lateral nodes with a short-axis of ≥7mm or ≥5mm with one or more malignant features (i.e. round shape, irregular margins, heterogeneity, loss of fatty hilum).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-06 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Lateral local recurrence | 3 years
  Lateral local recurrence diagnosed during the follow up

SECONDARY OUTCOMES:
Disease-free survival | 3 years
  The measure of time after treatment during which no sign of cancer is found.
Overall patient survival | 3 years
  The percentage of people who are alive 3 years after the surgery.
Morbidity and functional outcomes assessed by LARS questions | 3 years
  Use of questionnaire LARS
Quality of life as assessed by the EORTC QLQ-CR29 | 3 years
  Quality of life as assessed by the EORTC QLQ-CR29
Quality of life as assessed by the EQ-5D | 3 years
  Quality of life as assessed by the EQ-5D
Quality of life as assessed by the QLQ-C30 | 3 years
  Quality of life as assessed by the QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Miranda Kusters, MD, PhD, Principal Investigator — VUMedicalCentre
Locations (1):
- Amsterdam University Medical Centers, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
IPD data that underlie results in a publication can be made available upon reasonable request
Time Frame: Starting after initial publication of data
Access Criteria: Requests will be assessed by the study team

REFERENCES:
- [Result] Ogura A, Konishi T, Cunningham C, Garcia-Aguilar J, Iversen H, Toda S, Lee IK, Lee HX, Uehara K, Lee P, Putter H, van de Velde CJH, Beets GL, Rutten HJT, Kusters M; Lateral Node Study Consortium. Neoadjuvant (Chemo)radiotherapy With Total Mesorectal Excision Only Is Not Sufficient to Prevent Lateral Local Recurrence in Enlarged Nodes: Results of the Multicenter Lateral Node Study of Patients With Low cT3/4 Rectal Cancer. J Clin Oncol. 2019 Jan 1;37(1):33-43. doi: 10.1200/JCO.18.00032. Epub 2018 Nov 7. PMID 30403572
- [Result] Ogura A, Konishi T, Beets GL, Cunningham C, Garcia-Aguilar J, Iversen H, Toda S, Lee IK, Lee HX, Uehara K, Lee P, Putter H, van de Velde CJH, Rutten HJT, Tuynman JB, Kusters M; Lateral Node Study Consortium. Lateral Nodal Features on Restaging Magnetic Resonance Imaging Associated With Lateral Local Recurrence in Low Rectal Cancer After Neoadjuvant Chemoradiotherapy or Radiotherapy. JAMA Surg. 2019 Sep 1;154(9):e192172. doi: 10.1001/jamasurg.2019.2172. Epub 2019 Sep 18. PMID 31268504
- [Derived] van Geffen EGM, Sluckin TC, Hazen SJA, Horsthuis K, Intven M, van Dieren S, Beets G, Lange MM, Taggart MW, Beets-Tan RGH, Marijnen CAM, Konishi T, Tanis PJ, Kusters M; LaNoReC study group. Optimised treatment of patients with enlarged lateral lymph nodes in rectal cancer: protocol of an international, multicentre, prospective registration study after extensive multidisciplinary training (LaNoReC). BMJ Open. 2024 Oct 16;14(10):e083225. doi: 10.1136/bmjopen-2023-083225. PMID 39414276